CLINICAL TRIAL: NCT00545090
Title: An Open-label, Clinical Observation Extension Study to Assess Continuing Safety and Adherence in Patients With Postmenopausal Osteoporosis Receiving Monthly Oral Bonviva
Brief Title: ExBonAdAsia Study: A Study of Once Monthly Bonviva (Ibandronate) in Women With Post-Menopausal Osteoporosis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML19937
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Post Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ibandronate [Bonviva/Boniva]

INTERVENTIONS:
Drug: ibandronate [Bonviva/Boniva] — 150mg po monthly for 6 months

SUMMARY:
This single arm study will continue drug safety surveillance, and assessment of adherence, in patients with postmenopausal osteoporosis who have received monthly oral Bonviva in ML19930, the BonAdAsia study. All patients completing 6 months in ML19930 will continue to receive Bonviva (150mg po, monthly) for an additional 6 months. The anticipated time on study treatment is 3-12 months, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* patients responding to oral monthly Bonviva during the BonAdAsia study;
* willing to continue Bonviva treatment for a further 6 months.

Exclusion Criteria:

* none specified.

Max Age: 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2006-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
SAEs, AEs including fractures, adherence to treatment, clinical improvement, osteoporosis symptoms | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- Hong Kong, Hong Kong
- Indonesia (3):
  - Jakarta
  - Makassar
  - Surabaya
- Philippines (2):
  - Manila
  - Quezon City
- Taiwan (5):
  - Changhua
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Khon Kaen